CLINICAL TRIAL: NCT00373477
Title: A Randomized Trial of the Cost Effectiveness of Generalist Care Managers for the Treatment of Depression in Medicaid Recipients
Brief Title: A Study of the Cost Effectiveness of Generalist Care Managers for Depression Treatment in Medicaid Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Organization: University of North Carolina, Chapel Hill (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-fam/med-161; RWJF ID number: 048128
Record Dates: First submitted 2006-09-06; First posted 2006-09-08 (Estimated); Last update posted 2006-09-08 (Estimated); Status verified 2006-09

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Primary Care; Care Manager
MeSH Terms: conditions — Depressive Disorder, Major; Depression

INTERVENTIONS:
Procedure: Generalist Care Manager vs Usual Care

SUMMARY:
This project will enable the investigators to conduct a randomized clinical trial to demonstrate the value of generalist care managers in the treatment of depression in Medicaid patients seen in primary health care practices. Depressed patients will be recruited at two primary care practices in Western North Carolina and randomly assigned to either generalist care management or usual care. Patients in each condition will be assessed at baseline and six months follow-up. Outcomes will include depressive symptoms, level of functioning, and cost-effectiveness measures.

DETAILED DESCRIPTION:
Randomized trial among depressed Medicaid patients aged 18 years and older in 2 primary care practices in Western NC comparing an intervention with a GCM to usual care (UC) between July 2003 and February 2005. GCMs, already providing diabetes and asthma services, were further trained and given ongoing supervision to provide algorithm-based depression care to enhance guideline concordant treatment. GCMs provided elements of self-management, decision support, use of information systems, and core care management components.

ELIGIBILITY:
Inclusion Criteria:

* scoring 10 or greater on PHQ-9 and primary care physician verification of major depression by clinical exam; and
* willing to begin or continue antidepressant medication

Exclusion Criteria:

* bipolar disorder, psychotic symptoms, or active suicidal ideation requiring psychiatric admission (

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2003-07; Study Completion 2005-02

PRIMARY OUTCOMES:
Baseline, 3 and 6-month Patient Health Questionnaire (PHQ9) scores

SECONDARY OUTCOMES:
Baseline and 6-month Short Form (SF)-12 scores, Medicaid claims data; patient perception of treatment by self-report; review of GCM case notes, physician and office staff time study; physician and office staff focus groups

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Landis, MD, MPH, Principal Investigator — University of North Carolina
Locations (2):
- United States (2):
  - Mountain Area Health Education Center (MAHEC), Asheville, North Carolina
  - Hot Springs Health Program, Marshall, North Carolina